CLINICAL TRIAL: NCT01533857
Title: Pharmacokinetic Behavior of Phenolic Acids Derived From Black Tea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FDS-BNH-0379
Record Dates: First submitted 2012-02-05; First posted 2012-02-15 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2012-11

CONDITIONS: Cardiovascular Diseases
Keywords: Black tea; phenolic acids
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black tea (Experimental): black tea
  Interventions: Dietary Supplement: Black tea and phenolic acids
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: hot water

INTERVENTIONS:
Dietary Supplement: hot water — Hot water and placebo capsule
  Arms: placebo
Dietary Supplement: Black tea and phenolic acids — Black tea extract and capsule with phenolic acids
  Arms: Black tea

SUMMARY:
This study is set up to determine pharmacokinetics of phenolic acids after a single oral dose to healthy males.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* not smoking

Exclusion Criteria:

* use of NSAIDS and/or antibiotics
* no blood donation 1 months prior to screening

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of selected phenolic acids | up to 30 hrs

SECONDARY OUTCOMES:
plasma concentration of selected flavonoid metabolites | up to 30 hrs
Identification of unknown phenolic acids (metabolites of black tea) in plasma | up to 30 hrs
  It is still largely unknown which metabolites are formed in-vivo after black tea ingestions and circulating in human plasma. Untargeted profiling using LC-MS of plasma samples will be used to identify yet unknown polyphenols / phenolics and their conjugates in plasma and thus extent the hit-list of known metabolites in circulation after black tea consumption

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Optimed Eurofins, Gières, France

REFERENCES:
- [Derived] van Duynhoven J, van der Hooft JJ, van Dorsten FA, Peters S, Foltz M, Gomez-Roldan V, Vervoort J, de Vos RC, Jacobs DM. Rapid and sustained systemic circulation of conjugated gut microbial catabolites after single-dose black tea extract consumption. J Proteome Res. 2014 May 2;13(5):2668-78. doi: 10.1021/pr5001253. Epub 2014 Apr 10. PMID 24673575